CLINICAL TRIAL: NCT06629181
Title: The Effect of Educational Intervention on Digital Health Service Use in the Elderly on E-Health Literacy and Health Seeking Behavior: Randomized Controlled Study
Brief Title: E-Health Literacy and Health Seeking Behavior in the Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Zeynep Sacikara, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 16979
Record Dates: First submitted 2024-10-02; First posted 2024-10-08 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Health Services, Geriatric
Keywords: Digital Healthcare Service; elderly; eHealth Literacy; Health-seeking behavior
MeSH Terms: conditions — Health Behavior | interventions — Educational Status

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Elderly people will continue to receive routine care at the family health center.
- Intervention (Experimental): The group in which the intervention was made
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — The researchers will conduct a 4-week intervention for the intervention group participants.
  Technology Use Basic Information Training, MHRS and e-pulse Systems Usage Training Health literacy, mobile health application usage training Counseling Applications will be made at the end of the training
  Arms: Intervention

SUMMARY:
The purpose of this clinical trial is to determine the effect of an educational intervention on the use of digital health services for elderly individuals on e-health literacy and health seeking behavior.

The main questions it aims to answer are:

H 0 : There is no difference in terms of the total score of the e-health literacy scale.

H 0 : There is no difference in terms of the total score of the health seeking behavior scale.

The control group will continue their routine life. The researchers will conduct a 4-week intervention for the intervention group participants.

Technology Use Basic Information Training, MHRS and e-pulse Systems Usage Training Health literacy, mobile health application usage training Counseling Applications will be made at the end of the training.

DETAILED DESCRIPTION:
Electronic health (eHealth) is the use of information and communication technology in support of health and health-related areas and is increasingly integrated into health resources and service delivery (WHO, 2019). The World Health Organization (WHO) also recognizes that digital technologies have the potential to accelerate the achievement of the Sustainable Development Goals by improving health services (WHO, 2021). However, not everyone has sufficient access or skills to use digital technology to benefit from the benefits of eHealth. This situation cannot be ignored, especially for the elderly, who are a vulnerable group (Chang et al., 2021). Elderly health and reducing health inequalities are important issues among the Sustainable Development Goals 2030 (UNDP, 2023). In order to minimize inequalities, it is very important for the individual to adapt to the innovations of the age and develop technology use skills. (Akyazı, 2018; Tuna Uysal, 2020).

The sample size was determined by Power analysis. The sample was calculated as 29 elderly individuals for each group with a power of 90%, with an effect size of 0.88 in an experimental study (Xie 2011). Considering the 10% loss probability for the study group, the sample was determined as 32 for each group (experimental and control). Before randomization, elderly individuals who meet the inclusion criteria will be given general information about the study, their informed consent will be obtained for participation in the study, and a pre-test will be administered. Then, the block randomization method will be used for randomization, and opaque envelopes will be given by an independent researcher to conceal the assignment.

At the end of the study, the training given to the experimental group will also be given to the control group.

ELIGIBILITY:
Inclusion Criteria:

At least literate Having a smart phone Elderly individuals aged 60 and over Having internet access at home or at work

Exclusion Criteria:

Illiterate Not having a smart phone Individuals under the age of 60 Not having internet access at home or at work

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-10-07 (Actual); Primary Completion 2024-11-05 (Actual); Study Completion 2024-12-10 (Actual)

PRIMARY OUTCOMES:
Total score of e-health literacy scale | pre-test in the first meeting, posttest 4 weeks after registration
  There are 8 items measuring users&#39; knowledge, comfort and perceived skills in finding, evaluating and applying electronic health information regarding e-health problems. A 5-point Likert-type measurement is used to evaluate the items. The total score varies between 8 and 40, and higher scores indicate higher perceived skills in finding, evaluating and applying e-health information to make health decisions.

SECONDARY OUTCOMES:
Health Seeking Behavior Scale total score | pre-test in the first meeting, posttest 4 weeks after registration
  The scale consists of 3 dimensions and 12 items: online health seeking (6 items), professional health seeking (3 items), and traditional health seeking (3 items). The items in the scale were measured with 5-point Likert-type scale options (1 = strongly disagree, 5 = strongly agree). The minimum and maximum scores that can be obtained from the scale are 12 and 60, respectively. Higher scores represent better health seeking behavior.

CONTACTS AND LOCATIONS:
Overall Officials: ZEYNEP SAÇIKARA, Principal Investigator — https://www.erbakan.edu.tr/hemsirelikfak
Locations (1):
- Necmettin Erbakan Üniversitesi, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No